CLINICAL TRIAL: NCT03663777
Title: Effects of 12 Weeks of Isometric Handgrip Training in Blood Pressure in Patients With Peripheral Artery Disease
Brief Title: Handgrip Training in Patients With Peripheral Artery Disease
Acronym: Isopress_03
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Collaborators: Hospital Israelita Albert Einstein (Other)
Responsible Party: Principal Investigator, Raphael Mendes Ritti Dias, Professor, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ISO003
Record Dates: First submitted 2018-09-05; First posted 2018-09-10 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Isometric Handgrip Training (Experimental): Experimental group will perform home-based bilaterall handgrip exercise and will be recommended to increase daily physical activity levels.
  Interventions: Other: Isometric handgrip training
- Control group (Other): Control gorup will be recommended to increase daily physical activity level
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Isometric handgrip training — Intervention period will last 12 weeks. Experimental group will perform three sessions per week of home-based handgrip exercise. The exercise protocol will consist of eight sets of bilateral handgrip contraction of two minutes of isometric contraction, with 30% of maximum voluntary contraction, and two minutes of interval between sets. Patients will receive a diary to record the sessions and report difficulties during the training. The patients be recommended to increase daily physical activity levels, and weekly, there will be phone contacts with the patients to reinforce the exercise recommendations.
  Other Names: Isometric resistance exercise
  Arms: Isometric Handgrip Training
Other: Control Group — Intervention period will last 12 weeks. Patients will be recommended to increase daily physical activity levels, and weekly, there will be phone contacts to reinforce the recommendations.
  Arms: Control group

SUMMARY:
The aim of this study is to analyze the effects of isometric handgrip training (IHT) on blood pressure of hypertensive patients with peripheral arterial disease. Will be recruited 30 patients which will be randomized into 2 groups (15 per group), IHT and control group (CG). IHT group will training isometric contraction for 12 weeks. In CG patients will be encouraged to increase the level of physical activity. In the pre and post-intervention cardiovascular measures will be obtained.

DETAILED DESCRIPTION:
Meta-analyze studies have shown that 4 sets of 2 min of isometric handgrip training (IHT)reduces blood pressure (BP), reaching 10 mmHg for systolic and diastolic 7 mmHg in hypertensive patients after few weeks. However, using this protocol it was not observed any changes in BP in patients with peripheral artery disease. However, it is unknown whether reductions in BP does not occur after isometric handgrip training employing longer and protocol of IHT with more volume. The aim of this study is to analyze the effects of IHT on blood pressure of hypertensive patients with peripheral arterial disease. Will be recruited 30 patients, which will be randomized into 2 groups (15 per group), IHT and control group (CG). IHT group will hold three sessions per week with eight sets of two minutes of isometric contraction at 30% of maximal voluntary contraction and interval of two minutes between them, for 12 weeks. In the CG patients will be encouraged to increase the level of physical activity. In the pre and post-intervention, BP and cardiac autonomic modulationwill be assessed. Will be used to analyze two-factor variance for repeated measures, with group (IHT and CG) and the time (before and after 12 weeks) as factors and the post-hoc test of Newman-Keuls.

ELIGIBILITY:
Inclusion Criteria:

* Women in post-menopause phase without hormone replacement therapy
* Ankle-brachial index <0.90
* Not severe obese (≥ 35kg/m2)
* Not present amputation in the limbs
* Have blood pressure levels lower than 160mmHg for systolic and 105mmHg for diastolic

Exclusion Criteria:

* patients will only be excluded if they make any medication changes before completing the intervention period or present any health problems that prevent physical activity.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in blood pressure at 12 weeks | Baseline and 12 weeks
  Blood pressure will be measured before and after 12 weeks of intervention period on intervention and control group by an automatic blood pressure monitor (HEM-742, Omron Healthcare, Japan).

SECONDARY OUTCOMES:
Change from baseline in cardiac autonomic modulation at 12 weeks | Baseline and 12 weeks
  Cardiac autonomic modulation will be measured before and after 12 weeks of intervention period on intervention and control group by heart rate monitor (Polar, RS 800, USA).

CONTACTS AND LOCATIONS:
Overall Officials: Raphael Dias, PhD, Principal Investigator — University of Nove de Julho; Marilia Correia, PhD, Study Chair — University of Nove de Julho
Locations (2):
- Brazil (2):
  - Universidade Nove de Julho, São Paulo
  - Hospital Israelita Albert Einstein, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
WE plan to share the data upon requirement
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: After 1 year after the end of recruitment